CLINICAL TRIAL: NCT05370417
Title: Photobiomodulation and Glass Ionomer Sealant as Complementary Treatment for Hypersensitivity in Molars With MIH in Children - Protocol for a Blinded Randomized Clinical Trial.
Brief Title: Photobiomodulation and Glass Ionomer Sealant as Complementary Treatment for Hypersensitivity in Molars With MIH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBMDHMI
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hypomineralization Molar Incisor
MeSH Terms: conditions — Molar Hypomineralization | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The application of low-intensity laser will be simulated in one of the groups, to maintain the study blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Participants in this group received toothpaste with fluoride concentration ≥ 1000 ppm (Parts Per Million), glass ionomer sealant and simulated low-level laser.
  Interventions: Other: Use of fluoride toothpaste; Procedure: Simulated Laser Therapy; Procedure: Sealant application
- Study Group (Active Comparator): Participants in this group received toothpaste with fluoride concentration ≥ 1000 ppm (Parts Per Million), glass ionomer sealant and active low-level laser.
  Interventions: Other: Use of fluoride toothpaste; Radiation: Photobiomodulation; Procedure: Sealant application

INTERVENTIONS:
Other: Use of fluoride toothpaste — The participants received oral hygiene instructions - routine brushing twice per day with toothpaste containing 1000 ppm of fluoride. All participants received a toothbrush and toothpaste to ensure standardization. The aim of this intervention was to assess whether the participants' brushing technique would improve with desensitization.
Radiation: Photobiomodulation — For laser application, the following dosimetric parameters will be used:
  Low level laser diode (infra red) wavelength 808nm with a power of 100mW. Three sessions: initial session, after 48 hours and after one month. LLL was applied to three perpendicular points in contact with the surface on the mesial vestibular and distal cervical faces and in the center of the occlusal face. An energy of 1 J was applied for 10 seconds at each point.
  Arms: Study Group
Procedure: Simulated Laser Therapy — The same application described in the laser therapy group will be simulated, with the device turned off.
  Arms: Control Group
Procedure: Sealant application — A glass ionomer sealant will be applied to the occlusal surface of the first permanent molar.

SUMMARY:
Introduction: Photobiomodulation (PBM) shows promising results for the complementary treatment of dentin hypersensitivity; however, few studies have evaluated this treatment specifically for teeth affected by molar incisor hypomineralization (MIH). The aim of this study was to assess the effects of photobiomodulation combined with glass ionomer sealant on hypersensitivity in molars with MIH. Methods: Forty-nine children six to twelve years of age with a molar affected by MIH (Grade 3, 4a or 4b) of the MIH-TNI (Treatment Needs Index) criteria were randomly allocated to two groups - Group 1 (control group) (n = 25): toothpaste with fluoride concentration ≥ 1000 ppm (Parts Per Million) twice per day, glass ionomer sealant and simulated PBM; Group 2 (study group) (n = 24): toothpaste with fluoride concentration ≥ 1000 ppm twice per day, glass ionomer sealant and active PBM. Data collection involved the record of MIH, Schiff cold air sensitivity scale (SCASS), visual analog scale (VAS), the simplified oral hygiene index (OHI) and the colour, coverage, caries (CCC) sealant evaluation system. Results: Forty-six children completed the study and were evaluated one month after the onset of treatment. A significant reduction in the Schiff Cold Air Sensitivity Scale (SCASS) was found only in the active PBM group. Reductions in Visual Analog Scale (VAS) scores were observed in both groups, with a statistically significant difference between the groups at the 48-hour and 1-month assessments following PBM application. Similarly, significant differences in the Oral Hygiene Index (OHI) were found only in the active PBM group when comparing baseline values to those after 48 hours and one month. A significant difference between the groups was noted for sealant durability at one month, with better scores in the active PBM group. Conclusion: The administration of photobiomodulation combined with glass ionomer cement improves hypersensitivity and oral hygiene in molars with MIH. The improvement in oral hygiene increases the quantity of remaining sealant on teeth with MIH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (ASA I);
* Children aged 6 to 12 years with at least one permanent first molar affected by MIH grades 3 and 4 (a and b) according to the MIH Treatment Needs Index (TNI), and with hypersensitivity score 2 or higher on the visual analog scale (VAS);
* Molars with fractures and without pulp involvement or active caries;
* Molars with eruption of the entire occlusal surface and at least one-third of the vestibular surface.

Exclusion Criteria:

* Molars with hypersensitivity caused by carious lesions were excluded to avoid diagnostic confusion with pulpitis;
* Teeth that had undergone desensitizing treatments in the previous three months, except for daily use toothpaste;
* Those with fixed orthodontic appliances; Patients who experienced discomfort during the hypersensitivity test, or those unable to tolerate the procedure were also excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Changes in pain - Visual analog scale (VAS) | Baseline, 48 hours after the procedures and 1 month after.
  The perception of pain in children was assessed using the Wong-Baker Faces Pain Rating Scale. This scale facilitates communication, allowing for a more accurate assessment of the pain reported by the child.
Changes in the Schiff Cold Air Sensitivity Scale (SCASS) | Baseline, 48 hours after the procedures and 1 month after.
  The (SCASS) will be used to assess subject response to this stimulus (0=no response to the stimulus; 1=no response to the stimulus, patient considers stimulus to be painful; 2= response to stimulus, patient moves from the stimulus; 3= response to the stimulus, patient moves from the stimulus and requests immediate discontinuation of the stimulus).

SECONDARY OUTCOMES:
Changes in the Simplified Oral Hygiene Index (Greene and Vermillion) | Baseline, 48 hours after the procedures and 1 month after.
  Analysis of soft plaque deposit:
  Code 0 = no deposits or pigmentation Code 1 = deposits covering less than 1/3 or presence of pigmentation Code 2 = deposits covering more than 1/3 but less than 2/3 Code 3 = deposits covering more than 2/3 of tooth surface
Sealant Assessment System | Baseline, 48 hours after the procedures and 1 month after.
  The retention of the sealant was evaluated after 1 month using the CCC Sealant Evaluation System. For statistical purposes, the following classification was considered: A: sealant present; B: Sealant present on 50% of fissure pattern but some missing; C: Sealant present on 50% of fissure pattern.; D: no sealant present.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Bussadori, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Fossati AL, Mandetta ARH, Sobral APT, Bruno LH, Viarengo NO, Sertaje MRF, Santos EM, Goncalves MLL, Mesquita-Ferrari RA, Fernandes KPS, Horliana ACRT, Motta LJ, Deana AM, Dos Santos-Pinto LAM, Bussadori SK. Randomized clinical trial of photobiomodulation and glass ionomer sealant for hypersensitivity in molar incisor hypomineralization. Sci Rep. 2025 Aug 29;15(1):31911. doi: 10.1038/s41598-025-17454-8. PMID 40883469
- [Derived] Fossati AL, Sobral APT, Hermida Bruno MLL, Viarengo NO, Sertaje MRF, Santos EM, Goncalves MLL, Ferrari RAM, Fernandes KPS, Horliana ACRT, Motta LJ, Bussadori SK. Photobiomodulation and glass ionomer sealant as complementary treatment for hypersensitivity in molar incisor hypomineralisation in children: protocol for a blinded randomised clinical trial. BMJ Open. 2023 Jun 14;13(6):e068102. doi: 10.1136/bmjopen-2022-068102. PMID 37316315